CLINICAL TRIAL: NCT01355055
Title: Influences of Catheter-based Renal Denervation on Central Sympathetic Nervous System Regulation in Refractory Hypertension
Brief Title: Sympathetic Activity and Renal Denervation
Acronym: ReD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: PD Dr. med. Karsten Heusser, Hannover Medical School
Other Study IDs: DE-MHH-ReD-EK5853
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary hypothesis:

Catheter-based renal denervation reduces central sympathetic activation in patients with refractory hypertension.

Secondary hypotheses:

1. The magnitude of the individual depressor response after catheter-based renal denervation depends on the extent of sympathoinhibition.
2. Both, the reduction in arterial pressure and in central sympathetic activation are sustained over time up to 24±3 months after catheter-based renal denervation.
3. Catheter-based renal denervation resets the sympathetic baroreflex to lower blood pressure values.

ELIGIBILITY:
Inclusion Criteria:

* Refractory hypertension (as defined by the WHO: poorly controlled hypertension (>140/90 mmHg) despite adequate doses of at least three antihypertensive drugs including a diuretic)
* Men or women aged >18 years
* Intact peroneal nerve
* Written informed consent

Exclusion Criteria:

* Diseases, dysfunctions, or medications (such as NET inhibitors) that exclude a participation in the study according to the investigator.
* Legal incompetence or circumstances that interfere with the patient´s ability to fully understand scope, relevance, and/or consequences of participation in this study.
* People in custody
* hypersensitivity to clonidine, phenylephrine, or nitroprusside-sodium
* sick sinus syndrome, second or third degree AV block, bradycardia < 50 bpm (contraindication for clonidine)
* endogenous depression (contraindication for clonidine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with refractory hypertension, in whom catheter-based renal denervation is indicated and who are scheduled for this procedure, will be recruited from the outpatient clinic.
Sampling Method: Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2011-03

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Derived] Brinkmann J, Heusser K, Schmidt BM, Menne J, Klein G, Bauersachs J, Haller H, Sweep FC, Diedrich A, Jordan J, Tank J. Catheter-based renal nerve ablation and centrally generated sympathetic activity in difficult-to-control hypertensive patients: prospective case series. Hypertension. 2012 Dec;60(6):1485-90. doi: 10.1161/HYPERTENSIONAHA.112.201186. Epub 2012 Oct 8. PMID 23045466